CLINICAL TRIAL: NCT05067790
Title: A Phase 3b Study to Evaluate Higher Dose Nusinersen (BIIB058) in Patients With Spinal Muscular Atrophy Previously Treated With Risdiplam
Brief Title: A Study to Learn About the Effect of Higher Doses of Nusinersen (BIIB058) Given as Injections to Participants With Spinal Muscular Atrophy (SMA) Who Were Previously Treated With Risdiplam (ASCEND)
Acronym: ASCEND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 232SM303; 2021-001294-23 (EudraCT Number); 2023-505639-11 (Other: EU CTIS)
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Higher Dose Nusinersen (Experimental): All participants in the core study period, previously treated with risdiplam (nusinersen-naive participants and nusinersen-experienced participants), will receive HD nusinersen, administered as 2 loading doses of 50 milligrams (mg) each, approximately 2 weeks apart, followed by maintenance doses of 28 mg approximately every 4 months. Following the core study period, participants may be given the opportunity to receive maintenance doses of 28 mg nusinersen administered approximately every 4 months up to 2 years during the optional long-term extension (LTE) period.
  Interventions: Drug: Nusinersen

INTERVENTIONS:
Drug: Nusinersen — Administered as specified in the treatment arm
  Other Names: BIIB058; Spinraza

SUMMARY:
In this study, researchers will learn more about the use of a higher dose of nusinersen (BIIB058) in participants with spinal muscular atrophy (SMA). This study will focus on teenagers and adults who are unable to walk on their own and who have previously taken another drug for SMA called risdiplam.

The main goal of this study is to learn about the effect of high dose (HD) nusinersen on muscle and movement ability (motor function) in SMA. The main question that researchers want to answer is:

- How do the scores of a movement test called the Revised Upper Limb Module change from the start of treatment?

The Revised Upper Limb Module is a test used to measure a participant's ability to do specific tasks that involve their shoulders, arms, wrist, elbows, and hands. It measures the changes in their abilities over time.

Researchers will also learn more about the safety of HD nusinersen. They will check participants for adverse events and changes in vital signs, heart tests, and laboratory tests including blood and urine tests.

The study will be done as follows:

* Participants will be screened to check if they can join the study.
* After screening, participants will enter the Core Treatment period.
* At the start of the Core Treatment period, they will receive 2 "loading" doses of nusinersen. These are 50 mg doses of nusinersen given 2 weeks apart.
* Afterwards, they will continue to receive "maintenance" doses of nusinersen once every 4 months. These doses will be 28 mg.
* The Core Treatment period will last about 2 years, with a follow-up visit 4 months after the last dose.
* Participants who complete the Core Treatment period will have the option to continue receiving 28 mg of nusinersen in the Long-Term Extension (LTE) period for about 2 years. There will also be a follow-up visit 4 months after the last dose.
* Nusinersen will be given through a lumbar puncture, which involves injecting the drug into the fluid around the spinal cord in the lower back.
* In total, participants will have up to 18 study visits. They will also be called by researchers after each dose of nusinersen.
* Participants will stay in the study for about 4.5 years if they complete both the Core Treatment and LTE periods.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate motor function following treatment with HD nusinersen in participants with spinal muscular atrophy (SMA) previously treated with risdiplam.

The secondary objective of this study is to evaluate the safety and tolerability of HD nusinersen in participants with SMA previously treated with risdiplam.

ELIGIBILITY:
Key Inclusion Criteria:

* Genetic documentation of 5q SMA homozygous survival motor neuron-1 (SMN1) gene deletion or mutation or compound heterozygous mutation.
* Diagnosis of later-onset SMA with symptom onset at age >6 months.
* Aged ≥15 to ≤50 years at the time of informed consent
* Body weight >20 kg.
* Received oral risdiplam per the approved label or per the managed access program as follows

  1. Nusinersen-naive participants must have had prior treatment with risdiplam for ≥6 months before enrollment.
  2. Nusinersen-experienced participants must have stopped nusinersen for ≥16 months and must have been on risdiplam for ≥12 months before enrollment.
* Able to perform the age-appropriate functional assessments in the study.
* RULM entry item A score ≥3.
* RULM total score ≥5 and ≤30 at Screening.
* Nonambulatory, defined as not able to walk 15 feet (4.57 meters) independently without support.
* Willing to stop risdiplam treatment.
* Willing and able to start treatment with HD nusinersen.

Key Exclusion Criteria:

* Any major illness within 1 month before the screening examination or within 1 week prior to Screening and up to first dose administration.
* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy at any time during the Screening Period.
* Presence of an implanted shunt for the drainage of CSF or of an implanted central nervous system catheter.
* Permanent tracheostomy or permanent ventilation at Screening.
* The medical necessity, as defined by the Investigator, for noninvasive ventilation such as bilevel positive airway pressure or continuous positive airway pressure outside of regular sleep hours for any reason other than proactive SMA management, at Screening.
* History of bacterial meningitis, viral encephalitis, or hydrocephalus.
* Ongoing medical condition that according to the Investigator would interfere with the conduct and assessments of the study. An example is a medical disability (e.g., wasting or cachexia, severe anemia, and respiratory parameters) that would interfere with the assessment of safety or would compromise the ability of the participant to undergo study procedures.
* Participants who are pregnant or currently breastfeeding and those intending to become pregnant during the study.
* Treatment with an investigational drug, biological agent, or device within 30 days or 5 half-lives of the agent, whichever is longer, prior to Screening or anytime during the study; any prior or current treatment with gene therapy for the treatment of SMA.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2027-06-14 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
Change in Total Revised Upper Limb Module (RULM) Score | Up to Day 855
  The RULM is being utilized to assess upper limb functional abilities of participants with SMA. This test consists of upper limb performance items that are reflective of activities of daily living. The RULM is scored from 0 to 37 points, with higher scores indicating better function.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 1695
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death or in the view of the investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a birth defect, or is a medically important event.
Number of Participants With Change in Clinical Laboratory Parameters, Electrocardiogram (ECG), Vital Signs and Pulse Oximetry from Baseline | Up to Day 1695

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (43):
- United States (19):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Children's Hospital, Loma Linda, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Georgetown University, Washington D.C., District of Columbia
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - Memorial Healthcare, Owosso, Michigan
  - Columbia University, New York, New York
  - Wake Forest University - School of Medicine - Central, Winston-Salem, North Carolina
  - The Ohio State, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Neurology Rare Disease Center, Denton, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - FMUSP, São Paulo
- Germany (6):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen, Hesse
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Charité - Campus Virchow-Klinikum, Berlin
- Semmelweis Egyetem, Budapest, Hungary
- Italy (5):
  - Ospedale Pediatrico Bambino Gesù, Rome, Roma
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Fondazione Serena Onlus - Centro Clinico Nemo, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Ospedale S G Battista Molinette, Torino
- Japan (2):
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - NHO Osaka Toneyama Medical Center, Toyonaka-shi, Osaka
- Poland (4):
  - Szpital Specjalistyczny im. L.Rydygiera w Krakowie, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Spain (2):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- See also: Disclaimer: Residents in the United States may click here to find out more about participation in this trial. — https://www.ascendsmastudy.com/